CLINICAL TRIAL: NCT00297895
Title: A Phase III Multicenter Randomized Trial of Sentinel Lymphadenectomy and Complete Lymph Node Dissection Versus Sentinel Lymphadenectomy Alone in Cutaneous Melanoma Patients With Molecular or Histopathological Evidence of Metastases in the Sentinel Node
Brief Title: Multicenter Selective Lymphadenectomy Trial II (MSLT-II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSLT-II; P01CA029605 (NIH); R01CA189163 (NIH); NCT00389571 (obsolete NCT alias)
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Melanoma
Keywords: sentinel lymph node dissection; complete lymph node dissection; surgical
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound observation + delayed CLND if recurrence detected (Active Comparator)
  Interventions: Procedure: Monitoring with nodal ultrasound
- CLND (Active Comparator)
  Interventions: Procedure: Completion Lymphadenectomy

INTERVENTIONS:
Procedure: Completion Lymphadenectomy — complete lymph node dissection of lymph node basin with positive node
  Arms: CLND
Procedure: Monitoring with nodal ultrasound — serial ultrasound monitoring of SLND positive basin. If recurrence detected, subject has CLND.
  Arms: Ultrasound observation + delayed CLND if recurrence detected

SUMMARY:
Subjects must be diagnosed with melanoma. All subjects receive sentinel lymphadenectomy. If the subject is sentinel node positive and meets study requirements, the subject is randomized to receive either (1) completion lymphadenectomy (2) observation with nodal ultrasound. Subjects are then followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Between 18 and 75 years of age.
3. Have a primary melanoma that is cutaneous (including head, neck, trunk, extremity, scalp, palm, sole, subungual skin tissues).
4. Have clear margins following WLE.
5. ECOG performance status 0-1.
6. Life expectancy of at least 10 years from the time of diagnosis, not considering the melanoma in question, as determined by the PI.
7. Willing to return to the MSLT-II center for follow up examinations and procedures as outlined in the protocol.
8. Randomization and/or CLND (as appropriate to randomization arm) must be completed no more than 120 days following the diagnostic biopsy of the primary melanoma.
9. Have a melanoma-related tumor-positive SN, determined by either of the following methods:

   1. Diagnosis of tumor-positive SN by MSLT-II center institutional pathologist by either H&E or IHC (using S-100, Mart-1, and HMB-45).
   2. Diagnosis of tumor-positive SN by RT-PCR analysis performed at JWCI, provided the primary melanoma fits into one of the following categories:

      * Breslow thickness of 1.20 mm or greater and Clark Level III
      * Clark Level IV or V, regardless of Breslow thickness
      * Ulceration, regardless of Breslow thickness or Clark level

Exclusion Criteria:

1. History of previous or concurrent (i.e., second primary) invasive melanoma.
2. Primary melanoma of the eye, ears, mucous membranes or internal viscera. (Primary of the skin of the external ear is acceptable.)
3. Physical, clinical, radiographic or pathologic evidence of satellite, in-transit, regional, or distant metastatic disease.
4. Any additional solid tumor or hematologic malignancy during the past 5 years except T1 skin lesions of squamous cell carcinoma, basal cell carcinoma, or uterine cervical cancer.
5. Skin grafts, tissue transfers or flaps that have the potential to alter the lymphatic drainage pattern from the primary melanoma to a LN basin.
6. Allergy to vital blue dye or any radiocolloid.
7. Inability to localize 1-2 SN drainage basins via LM (e.g., no basins found, more than 2 basins found, proximity of the primary melanoma to the regional draining basin, etc.)
8. CLNDs or SLs (before evaluation of the current melanoma) that may have altered the lymphatic drainage pattern from the primary cutaneous melanoma to a potential LN basin.
9. Organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the full protocol, or be exacerbated by therapy (e.g., severe depression).
10. Melanoma-related operative procedures not corresponding to criteria described in the protocol.
11. Primary or secondary immune deficiencies or known significant autoimmune disease.
12. History of organ transplantation.
13. Oral or parenteral immunosuppressive agents (not topical or inhaled steroids) at any time during study participation or within 6 months prior to enrollment.
14. Pregnant or lactating women.
15. Participation in concurrent therapy protocols of alternative local nodal basin therapies that might confound the analysis of this trial is not permitted. For example, radiation of a non-resected node basin is not acceptable because it might influence outgrowth of residual melanoma in that nodal basin. However, systemic adjuvant therapy or clinical trial adjuvant protocols after the finding of a positive node on LM/SL or delayed nodal recurrence in the ultrasound observation arm are both acceptable according to the standard of care at the multicenter site. Patients with positive sentinel nodes or thick primary melanomas who are considered by the multicenter site's investigator as high-risk may receive systemic adjuvant therapy according to the standard practice of that particular site.
16. SLND pathology shows, on microscopic examination, that melanoma extends through the lymph node capsule into the adjacent soft tissue.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1939 (Actual)
Dates: Start 2004-09-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Melanoma-specific survival. This is defined as the time between the date of a subject's randomization (or date of CLND for those randomized to the CLND arm) and the date of death due to melanoma. Subjects are followed until death or 10yrs. | 10 years

SECONDARY OUTCOMES:
Disease-free survival over 10 years of follow up | 10 years
Recurrence during 10 years of follow up | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Essner, M.D., Principal Investigator — Saint John's Cancer Institute
Locations (63):
- United States (39):
  - Sharp Hospital, San Diego, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Memorial Hospital - Colorado Springs, Colorado Springs, Colorado
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - St. Louis University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Buffalo General Hospital, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Feinstein Institute for Medical Research, Great Neck, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SUNY at Stony Brook Hospital Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Pennsylvania State Hershey Cancer Institute, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Main Line Surgeons, Wynnewood, Pennsylvania
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Dallas Surgical Group, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - IHC Cancer Services Intermountain Medical Center, Salt Lake City, Utah
  - Hunstman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Careplex Hospital, Newport News, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (5):
  - Newcastle Melanoma Unit, Newcastle, New South Wales
  - Melanoma Institute Australia, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Alfred Hospital, East Hawthorn, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Sunnybrook Health Sciences Center, Toronto, Ontario
- Helsinki Unversity Hospital, Helsinki, Finland
- Germany (3):
  - U. Hosp. Schleswig-Holstein/Campus Lubeck, Lübeck
  - City Hospital of Nurnberg, Nuremberg
  - University of Wurzburg, Würzburg
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (4):
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale dei Tumori Napoli, Naples
  - Istituto Oncologico Veneto - University of Padova, Padua
  - Padua University - Clinica Chirurgica II, Padua
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Hospital Clinic Barcelona, Barcelona, Spain
- Swedish Melanoma Study Group, Lund, Sweden
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University of Zurich, Zurich
- United Kingdom (2):
  - Norfolk and Norwich University Hospital, Norfolk, Norwich
  - Saint Thomas's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Multicenter Selective Lymphadenectomy Trials Study Group; Crystal JS, Thompson JF, Hyngstrom J, Caraco C, Zager JS, Jahkola T, Bowles TL, Pennacchioli E, Beitsch PD, Hoekstra HJ, Moncrieff M, Ingvar C, van Akkooi A, Sabel MS, Levine EA, Agnese D, Henderson M, Dummer R, Neves RI, Rossi CR, Kane JM 3rd, Trocha S, Wright F, Byrd DR, Matter M, Hsueh EC, MacKenzie-Ross A, Kelley M, Terheyden P, Huston TL, Wayne JD, Neuman H, Smithers BM, Ariyan CE, Desai D, Gershenwald JE, Schneebaum S, Gesierich A, Jacobs LK, Lewis JM, McMasters KM, O'Donoghue C, van der Westhuizen A, Sardi A, Barth R, Barone R, McKinnon JG, Slingluff CL, Farma JM, Schultz E, Scheri RP, Vidal-Sicart S, Molina M, Testori AAE, Foshag LJ, Van Kreuningen L, Wang HJ, Sim MS, Scolyer RA, Elashoff DE, Cochran AJ, Faries MB. Therapeutic Value of Sentinel Lymph Node Biopsy in Patients With Melanoma: A Randomized Clinical Trial. JAMA Surg. 2022 Sep 1;157(9):835-842. doi: 10.1001/jamasurg.2022.2055. PMID 35921122
- [Derived] Faries MB, Thompson JF, Cochran AJ, Andtbacka RH, Mozzillo N, Zager JS, Jahkola T, Bowles TL, Testori A, Beitsch PD, Hoekstra HJ, Moncrieff M, Ingvar C, Wouters MWJM, Sabel MS, Levine EA, Agnese D, Henderson M, Dummer R, Rossi CR, Neves RI, Trocha SD, Wright F, Byrd DR, Matter M, Hsueh E, MacKenzie-Ross A, Johnson DB, Terheyden P, Berger AC, Huston TL, Wayne JD, Smithers BM, Neuman HB, Schneebaum S, Gershenwald JE, Ariyan CE, Desai DC, Jacobs L, McMasters KM, Gesierich A, Hersey P, Bines SD, Kane JM, Barth RJ, McKinnon G, Farma JM, Schultz E, Vidal-Sicart S, Hoefer RA, Lewis JM, Scheri R, Kelley MC, Nieweg OE, Noyes RD, Hoon DSB, Wang HJ, Elashoff DA, Elashoff RM. Completion Dissection or Observation for Sentinel-Node Metastasis in Melanoma. N Engl J Med. 2017 Jun 8;376(23):2211-2222. doi: 10.1056/NEJMoa1613210. PMID 28591523
- See also: John Wayne Cancer Institute Clinical Trials (sponsor) — https://www.saintjohnscancer.org/clinical-trials/

DOCUMENTS (1):
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT00297895/ICF_000.pdf